CLINICAL TRIAL: NCT01298401
Title: A Phase I Study of Induction AMG 479 and Gemcitabine, Followed by AMG 479, Capecitabine, and 3D-Conformal Radiation Therapy (3D-CRT) With Subsequent Maintenance Therapy for Locally Advanced Pancreatic Cancer
Brief Title: Ganitumab and Gemcitabine Hydrochloride Followed by Radiation Therapy, Ganitumab, Capecitabine, and Maintenance Therapy in Treating Patients With Locally Advanced Cancer of the Pancreas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 1102; CDR0000695567
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage IIB pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ganitumab; Capecitabine; Gemcitabine; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm A (Experimental): Dose level -1A (Ganitumab 6 mg/kg, Capecitabine 825mg/m2)
  Interventions: Biological: ganitumab; Drug: capecitabine; Drug: gemcitabine hydrochloride; Radiation: 3-dimensional conformal radiation therapy
- Arm B (Experimental): Dose level 1A (Ganitumab 12 mg/kg, Capecitabine 825mg/m2)
  Interventions: Biological: ganitumab; Drug: capecitabine; Drug: gemcitabine hydrochloride; Radiation: 3-dimensional conformal radiation therapy
- Arm C (Experimental): Dose level 2A (Ganitumab 20 mg/kg, Capecitabine 825mg/m2)
  Interventions: Biological: ganitumab; Drug: capecitabine; Drug: gemcitabine hydrochloride; Radiation: 3-dimensional conformal radiation therapy
- Arm D (Experimental): Dose level -1B (Ganitumab 6 mg/kg, Capecitabine 625mg/m2)
  Interventions: Biological: ganitumab; Drug: capecitabine; Drug: gemcitabine hydrochloride; Radiation: 3-dimensional conformal radiation therapy
- Arm E (Experimental): Dose level 1B (Ganitumab 12 mg/kg, Capecitabine 625mg/m2)
  Interventions: Biological: ganitumab; Drug: capecitabine; Drug: gemcitabine hydrochloride; Radiation: 3-dimensional conformal radiation therapy
- Arm F (Experimental): Dose level 2B (Ganitumab 20 mg/kg, Capecitabine 625mg/m2)
  Interventions: Biological: ganitumab; Drug: capecitabine; Drug: gemcitabine hydrochloride; Radiation: 3-dimensional conformal radiation therapy

INTERVENTIONS:
Biological: ganitumab
Drug: capecitabine
Drug: gemcitabine hydrochloride
Radiation: 3-dimensional conformal radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as ganitumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as gemcitabine hydrochloride and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Specialized radiation therapy, such as 3-dimensional conformal radiation therapy, that delivers a high-dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase I trial is studying the side effects and best dose of ganitumab when given together with gemcitabine hydrochloride followed by radiation therapy, ganitumab, capecitabine, and maintenance therapy in treating patients with locally advanced cancer of the pancreas.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the maximum dose of ganitumab, up to a target dose of 20 mg/kg, given concurrently with capecitabine and radiotherapy following induction ganitumab and gemcitabine hydrochloride in patients with locally advanced pancreatic cancer.

Secondary

* To evaluate the safety profile of induction therapy comprising ganitumab and gemcitabine hydrochloride, followed by ganitumab and concurrent chemoradiation, and subsequently by maintenance ganitumab and gemcitabine hydrochloride until disease progression in patients with locally advanced pancreatic cancer.
* To evaluate response and overall survival of patients treated at the maximum dose of ganitumab given concurrently with capecitabine and radiotherapy following induction ganitumab and subsequently followed by maintenance ganitumab and gemcitabine hydrochloride until disease progression.

OUTLINE: This is a multicenter, dose-escalation study of ganitumab followed by an expanded cohort study.

Induction therapy: Patients receive ganitumab IV over 1-2 hours on days 1 and 15 and gemcitabine hydrochloride IV over 30 minutes on days 1, 15, and 22. Treatment repeats every 28 days for 2 courses.

Concurrent therapy: Beginning 10-28 days later, patients undergo 3-dimensional conformal radiotherapy once daily, 5 days a week for 5.5 weeks beginning on day 1. Patients also receive concurrent ganitumab IV over 1-2 hours on days 1, 15, and 29 and capecitabine orally (PO) twice daily on days 1-5 weekly for 5.5 weeks.

Maintenance therapy: Beginning 21-42 days later, patients receive ganitumab IV over 1-2 hours on days 1 and 15 and gemcitabine hydrochloride IV over 30 minutes on days 1, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years, every 4 months for 1 year, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed (histologic or cytologic) locally advanced adenocarcinoma of the pancreas

  * Patients must have unresectable disease based on institutional standardized criteria of unresectability or medical inoperability
* Patients with or without regional adenopathy are eligible
* No distant metastases based upon the following minimum diagnostic workup:

  * History and/or physical examination, including collection of weight and vital signs, within 28 days prior to study entry
  * Abdominal and/or pelvic CT scan with IV contrast or MRI scan within 21 days prior to study entry
  * Chest CT scan or whole-body PET/CT within 21 days prior to study entry
* No second malignancy or peritoneal seeding

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin (Hgb) ≥ 10.0 g/dL (the use of transfusion or other intervention to achieve Hgb ≥ 10.0 g/dL is acceptable)
* Glycosylated hemoglobin (HgbA1c) ≤ 8%
* Serum creatinine ≤ 1.5 mg/dL
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 3 times upper limit of normal (ULN)
* Total bilirubin < 3.0 mg/dL
* Alkaline phosphatase < 3 times ULN
* Fasting blood glucose < 160 mg/dL

  * Patients with a non-fasting blood glucose > 160 mg/dL (8.9 mmol/L) must have a fasting blood glucose ≤ 160 mg/dL (8.9 mmol/L) in order to be eligible
* No grade 2 or worse hearing impairment
* Negative serum pregnancy test (if applicable)
* Women of childbearing potential and men who are sexually active must be willing/able to use medically acceptable forms of contraception during the course of the study, and for 3 months (6 months for men) after the last study drug administration
* Not pregnant or nursing
* Ability to swallow oral medications
* At least 3 years since prior malignancy except non-melanomatous skin cancer or carcinoma in situ of the breast, oral cavity, or cervix
* No severe active co-morbidity, defined as any of the following:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within 6 months prior to study entry
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization, or precluding study therapy within 30 days before registration
  * Uncontrolled malabsorption syndrome significantly affecting gastrointestinal function
  * Any unresolved bowel or bile duct obstruction
  * Major resection of the stomach or small bowel that could affect the absorption of capecitabine
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition

    * HIV testing is not required for entry into this protocol
  * Existing venous thromboembolism requiring anti-coagulation therapy
* No prior allergic reaction to capecitabine or gemcitabine hydrochloride

PRIOR CONCURRENT THERAPY:

* No prior systemic chemotherapy for pancreatic cancer

  * Prior chemotherapy for malignancies other than pancreatic cancer is allowed provided chemotherapy was completed > 3 years prior to study entry
* No prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* More than 28 days since any prior major surgery

  * Insertion of a vascular access device, insertion of a biliary stent, exploratory laparotomy, or laparoscopy are not considered major surgery
* No prior ganitumab
* Patients requiring concurrent oral anticoagulants (e.g., Coumadin, warfarin) are eligible provided there is increased vigilance with respect to monitoring international normalized ratio (INR)
* No concurrent participation in another clinical treatment trial
* No concurrent intensity-modulated radiotherapy
* No other concurrent therapy including the following:

  * Other investigational or approved chemotherapeutic agents
  * Other monoclonal antibody
  * Sorivudine or brivudine A
  * Cimetidine
  * G-CSF agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity of ganitumab and capecitabine given concurrently with radiotherapy | From start of chemoradiation to 21 days after the end of chemoradiation

SECONDARY OUTCOMES:
Response rate (for patients treated at maximum-tolerated dose of ganitumab) | Analysis occurs after all patients have been potentially followed for 1 year
Overall survival (for patients treated at maximum-tolerated dose of ganitumab) | Analysis occurs after all patients have been potentially followed for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H. Crane, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (10):
- United States (10):
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Northmain Radiation Oncology, Providence, Rhode Island
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas